CLINICAL TRIAL: NCT03454685
Title: The Role of Microbiota on the Development of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 745435
Record Dates: First submitted 2018-01-21; First posted 2018-03-06 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: NSCLC, Stage I; NSCLC, Stage II; NSCLC, Stage III; NSCLC Stage IV; Healthy Subjects
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — We intend to collect the following samples：
  1. Blood samples
  2. Stool samples
  3. Sputum samples
  4. Tumor tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NCSLC group: NSCLC patients,including stage I to stage IV.
  Interventions: Other: without intervention type
- Healthy subjects: healthy subjects
  Interventions: Other: without intervention type

INTERVENTIONS:
Other: without intervention type — Without intervention,this study is just an observational study.

SUMMARY:
Relationship between human microbiota and epidemiology of lung cancer

DETAILED DESCRIPTION:
In this study,We aim to find some kinds of human microbiota , which were associated with development of non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer patients

Exclusion Criteria:

* long-term workers in the polluted environment, Patients who had used antibiotics within 1 month before sampling,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Just confirmed non-small cell lung cancer patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Relationship Between Human Microbiota and Epidemiology of Lung Cancer | 1 year
  Find some human microbes that are associated with the development of lung cancer, we can detect these human microbiological content as a biomarker of lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: dong xiaorong, Dr, Study Director — china government
Locations (1):
- Union hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Lu H, Gao NL, Tong F, Wang J, Li H, Zhang R, Ma H, Yang N, Zhang Y, Wang Y, Liang Z, Zeng H, Chen WH, Dong X. Alterations of the Human Lung and Gut Microbiomes in Non-Small Cell Lung Carcinomas and Distant Metastasis. Microbiol Spectr. 2021 Dec 22;9(3):e0080221. doi: 10.1128/Spectrum.00802-21. Epub 2021 Nov 17. PMID 34787462